CLINICAL TRIAL: NCT06599892
Title: Rethinking CF Organization of Care in the Era of Highly Effective Modulator: a Nationwide Research Program HORIZON.
Brief Title: CF Organization of Care in the Era of Highly Effective Modulator.
Acronym: HORIZON
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0749
Record Dates: First submitted 2024-08-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic; organisation; relationship; intervention; healthcare; mapping; fibrosis
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients from the 47 CF French center: National registry indicator study = 7513 patients in total, including 5000 eligible for highly effective CFTRm, for the study of pathways at national level, for which clinical and healthcare consumption data are available in the national registry linked to the SNDS
  Interventions: Other: Intervention mapping
- Healthcare professionels: Case study: 8 to 10 CRCMs, 7 to 8 professionals and 7 to 8 patients per CRCM, i.e. 56 to 80 professionals, 200 to 400 patients DELPHI: panel of 80 professionals and patients/parents
  Interventions: Other: Intervention mapping

INTERVENTIONS:
Other: Intervention mapping — Intervention mapping is a model combining patient and professional questionnaires and a qualitative survey using individual interviews with patients and focus groups with professionals to identify the obstacles and levers to change at the level of patients, professionals and organisations.

SUMMARY:
Recently, triple therapy has made it possible to extend access to these modulators to a large proportion of the patient population, with spectacular clinical benefits, provided the patient carries at least one F508del mutation.

The hypothesis is that the arrival of CFTRmHEs has considerably altered the way cystic fibrosis is managed, requiring a rethink of how the CRCMs are organised, and a redefinition of the practices and missions of professionals, as well as the patient-professional relationship.

DETAILED DESCRIPTION:
The organisation of cystic fibrosis care in France, within the Muco-CFTR rare disease network, is based on 47 cystic fibrosis resource and competence centres (CRCMs), which bring together multidisciplinary resources (doctors, physiotherapists, nurses, psychologists, dieticians, social workers) to ensure the continuity and coordination of patients' care pathways, taking into account the physical, psychological, educational/professional and social consequences of the disease. The CRCMs' missions are based on the National Diagnosis and Care Protocol (PNDS 2017). The recent arrival of highly effective CFTR modulators (CFTRmHE) in the arsenal of treatments is a therapeutic revolution for 83% of patients in the French Cystic Fibrosis Registry who are eligible for this treatment. Recently, triple therapy has made it possible to extend access to these modulators to a large proportion of the patient population, with spectacular clinical benefits, provided the patient carries at least one F508del mutation. This treatment improves lung function and body mass index, and reduces pulmonary exacerbations, with good tolerability. These results have led to its approval in 2019 in the United States and 2020 in Europe. Real-life results from 245 patients confirmed a spectacular improvement in respiratory function and nutritional status, to the extent that the indication for lung transplantation was suspended in 47 of the 53 patients concerned. The majority of eligible patients started treatment in 2021. The clinical benefits have prompted some patients to abandon standard treatments (respiratory physiotherapy, bronchial fluidisers) and to reconsider the way they are managed at the CRCM (spacing of visits, teleconsultation). However, in the absence of hindsight, it is not possible at present to make recommendations on reducing the burden of care.

The hypothesis is that the arrival of CFTRmHEs has considerably altered the way cystic fibrosis is managed, requiring a rethink of how the CRCMs are organised, and a redefinition of the practices and missions of professionals, as well as the patient-professional relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 and over with cystic fibrosis treated with CFTRmHE for at least 12 months
* Patients aged over 6 years with cystic fibrosis not eligible for CFTRmHE treatment
* Families of patients under 18 years of age
* Professionals working in a CRCM for more than 12 months, physiotherapists and community nurses involved in the management of cystic fibrosis.

Exclusion Criteria * :

* Refusal to participate
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In each phase we will use the sample size recommendations for each methodological approach
  * National surveys by CRCM questionnaire: all national CRCM centres will be contacted by the network.
  * National registry indicator study = 7513 patients in total, including 5000 eligible for highly effective CFTRm, for the study of pathways at national level, for which clinical and healthcare consumption data are available in the national registry linked to the SNDS.
  * Case study: 8 to 10 CRCMs, 7 to 8 professionals and 7 to 8 patients per CRCM, i.e. 56 to 80 professionals, 56 to 80 patients.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Obtaining a national consensus on a proposal for a new organisation of the cystic fibrosis care pathway, including the CRCMs and the liberal network | The outcome measure will be measured at the twelfth month of the survey.
  It will be measured by a mixed approach based on the intervention mapping model combining patient and professional questionnaires and a qualitative survey using individual interviews with patients and focus groups with professionals to identify the obstacles and levers to change at the level of patients, professionals and organisations.
  The main outcome measure is to establish a new organization of care for pwCF and HCPs in the era of HEMT by the develop an evaluation plan using a community-based participatory approach to promote external validity.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe REIX, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Groupement Hospitalier Est Pediatric CFcenter, Lyon, France

IPD SHARING:
Plan to Share IPD: No